CLINICAL TRIAL: NCT00484705
Title: Polycystic Ovary Syndrome (PCOS) - The Female Metabolic Syndrome Genes And Processes In The Aetiology And Pathogenesis Of PCOS And Identification Of New Treatment Strategies
Brief Title: Polycystic Ovary Syndrome (PCOS) - Effect Of Physical Exercise And Electroacupuncture
Acronym: PCOSNTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: VGFOUREG-7861; K2005-72VP-15445-01A; K2005-72VX-15276-01AK; LUA/ALF7092; DIA2006-001; Novo Nordisk Foundation
Record Dates: First submitted 2007-06-08; First posted 2007-06-11 (Estimated); Last update posted 2009-11-10 (Estimated); Status verified 2009-11

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Androgens; Menstrual pattern; Insulin resistance; Adipocytes; Obesity; Stress; Muscle sympathetic nerve activity; Psychological distress and quality of life
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance; Obesity | interventions — Electroacupuncture; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low-frequency electro-acupuncture (Experimental)
  Interventions: Procedure: Electroacupuncture
- Physical exercise (Experimental)
  Interventions: Procedure: Physical exercise
- Untreated control (Active Comparator)
  Interventions: Procedure: Untreated control

INTERVENTIONS:
Procedure: Electroacupuncture
  Arms: Low-frequency electro-acupuncture
Procedure: Physical exercise
  Arms: Physical exercise
Procedure: Untreated control
  Arms: Untreated control

SUMMARY:
Hypothesis:

The overall hypothesis is that women with PCOS, both obese and non-obese, have larger adipocytes, altered metabolism and signs of inflammation in adipose tissue and that these changes are associated with high sympathetic nerve activity, hyperandrogenism hyperinsulinaemia, insulin resistance with progression to type II diabetes and cardiovascular disease (CVD) as well as psychological distress and reduced quality of life. Physical exercise and electro-acupuncture decrease high concentrations of androgens, induce regulare menstrual pattern, inhibits high sympathetic activity and restore the PCOS induced disturbances.

DETAILED DESCRIPTION:
Primary outcome: Changes in androgen concentrations and menstrual pattern

Secondary outcome: changes in sympathetic nerve activity, uterus peristalsis, ovarian morphology, adipose tissue related variables, insulin sensitivity, coagulation factors and health related quality of life and symptoms of anxiety and depression.

ELIGIBILITY:
Inclusion Criteria:

* To get the diagnosis polycystic ovary syndrome (PCOS), ultrasonography should reveal at least 1 ovary with PCO according to the Rotterdam diagnostic criteria as well as one of the following two symptoms:

  1. Anovulation/oligoovulation defined as ≥ 35 days during the last year
  2. Clinical signs of hyperandrogenism (hirsutism, acne)

Exclusion Criteria:

* Cardiovascular disease
* Diabetes mellitus
* Other endocrine disease (congenital adrenal hyperplasia, androgen producing tumour, Cushing's syndrome)
* Estrogen/gestagen treatment during the last 3 months
* Breast-feeding the last 6 months
* Antiandrogen treatment the last 3 months

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2005-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
To measure if physical exercise and electro-acupuncture restores endocrine, neuroendocrine, metabolic and immunological disturbances related to sympathetic nerve activity as well as psychological distress and improve quality of life in women with PCOS. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Elisabet Stener-Victorin, Prof, PhD, Principal Investigator — Sahlgrenska Academy, Göteborg University
Locations (1):
- Institute of Neuroscience and Physiology, Sahlgrenska Academy, Göteborg University, Gothenburg, Sweden

REFERENCES:
- [Derived] Leonhardt H, Hellstrom M, Gull B, Lind AK, Nilsson L, Janson PO, Stener-Victorin E. Ovarian morphology assessed by magnetic resonance imaging in women with and without polycystic ovary syndrome and associations with antimullerian hormone, free testosterone, and glucose disposal rate. Fertil Steril. 2014 Jun;101(6):1747-56.e1-3. doi: 10.1016/j.fertnstert.2014.02.022. Epub 2014 Mar 21. PMID 24661732
- [Derived] Leonhardt H, Gull B, Stener-Victorin E, Hellstrom M. Ovarian volume and antral follicle count assessed by MRI and transvaginal ultrasonography: a methodological study. Acta Radiol. 2014 Mar;55(2):248-56. doi: 10.1177/0284185113495835. Epub 2013 Aug 7. PMID 23926234
- [Derived] Stener-Victorin E, Holm G, Janson PO, Gustafson D, Waern M. Acupuncture and physical exercise for affective symptoms and health-related quality of life in polycystic ovary syndrome: secondary analysis from a randomized controlled trial. BMC Complement Altern Med. 2013 Jun 13;13:131. doi: 10.1186/1472-6882-13-131. PMID 23763822
- [Derived] Billhult A, Stener-Victorin E. Acupuncture with manual and low frequency electrical stimulation as experienced by women with polycystic ovary syndrome: a qualitative study. BMC Complement Altern Med. 2012 Apr 3;12:32. doi: 10.1186/1472-6882-12-32. PMID 22471422
- [Derived] Stener-Victorin E, Baghaei F, Holm G, Janson PO, Olivecrona G, Lonn M, Manneras-Holm L. Effects of acupuncture and exercise on insulin sensitivity, adipose tissue characteristics, and markers of coagulation and fibrinolysis in women with polycystic ovary syndrome: secondary analyses of a randomized controlled trial. Fertil Steril. 2012 Feb;97(2):501-8. doi: 10.1016/j.fertnstert.2011.11.010. Epub 2011 Dec 9. PMID 22154367
- [Derived] Manneras-Holm L, Baghaei F, Holm G, Janson PO, Ohlsson C, Lonn M, Stener-Victorin E. Coagulation and fibrinolytic disturbances in women with polycystic ovary syndrome. J Clin Endocrinol Metab. 2011 Apr;96(4):1068-76. doi: 10.1210/jc.2010-2279. Epub 2011 Jan 20. PMID 21252248
- [Derived] Manneras-Holm L, Leonhardt H, Kullberg J, Jennische E, Oden A, Holm G, Hellstrom M, Lonn L, Olivecrona G, Stener-Victorin E, Lonn M. Adipose tissue has aberrant morphology and function in PCOS: enlarged adipocytes and low serum adiponectin, but not circulating sex steroids, are strongly associated with insulin resistance. J Clin Endocrinol Metab. 2011 Feb;96(2):E304-11. doi: 10.1210/jc.2010-1290. Epub 2010 Nov 17. PMID 21084397
- [Derived] Jedel E, Labrie F, Oden A, Holm G, Nilsson L, Janson PO, Lind AK, Ohlsson C, Stener-Victorin E. Impact of electro-acupuncture and physical exercise on hyperandrogenism and oligo/amenorrhea in women with polycystic ovary syndrome: a randomized controlled trial. Am J Physiol Endocrinol Metab. 2011 Jan;300(1):E37-45. doi: 10.1152/ajpendo.00495.2010. Epub 2010 Oct 13. PMID 20943753